CLINICAL TRIAL: NCT05760976
Title: Median Effective Dose of Cisatracurium for the Prevention of Fasciculation Caused by the Injection of Succinylcholine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhuan Zhang, Director, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20230226
Record Dates: First submitted 2023-02-26; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Fasciculation; Succinylcholine
MeSH Terms: conditions — Fasciculation | interventions — cisatracurium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Age range of 18 to 44 years olds (Experimental): The initial dose of cisatracurium for pre-injection was set at 0.015mg/kg according to previous literature and preliminary test results. The dose of cisatracurium was according to the patients' fasciculation level. If there is no fasciculation (negative reaction), the dose of cisatracurium in the next patient will be reduced until the patient has fasciculation. If there is fasciculation (positive reaction), the dose of cisatracurium will be increased in the next patient until the patient has no fasciculation.
  Interventions: Drug: Cisatracurium
- Age range of 45 to 59 years olds (Experimental): The initial dose of cisatracurium for pre-injection was set at 0.015mg/kg according to previous literature and preliminary test results. The dose of cisatracurium was according to the patients' fasciculation level. If there is no fasciculation (negative reaction), the dose of cisatracurium in the next patient will be reduced until the patient has fasciculation. If there is fasciculation (positive reaction), the dose of cisatracurium will be increased in the next patient until the patient has no fasciculation.
  Interventions: Drug: Cisatracurium
- Age range of 60 to 80 years olds (Experimental): The initial dose of cisatracurium for pre-injection was set at 0.015mg/kg according to previous literature and preliminary test results. The dose of cisatracurium was according to the patients' fasciculation level. If there is no fasciculation (negative reaction), the dose of cisatracurium in the next patient will be reduced until the patient has fasciculation. If there is fasciculation (positive reaction), the dose of cisatracurium will be increased in the next patient until the patient has no fasciculation.
  Interventions: Drug: Cisatracurium

INTERVENTIONS:
Drug: Cisatracurium — Advanced intravenous injection of cisatracurium before the succinylcholine injection

SUMMARY:
Succinylcholine is currently the only depolarizing neuromuscular blocker widely used in anesthesia induction and is the drug of choice for rapid sequential anesthesia induction. However, with succinylcholine, varying degrees of muscle fibrillation and muscle pain occur. Intravenous injection of succinylcholine caused by myomuscular fibrillation can cause increased intragastric pressure, intraocular pressure and intracranial pressure, increased serum potassium and postoperative myalgia, increased the incidence of adverse events such as needle prolapse, extravasation of injected drugs, and reduced perioperative comfort of patients. Pretreatment with cisatracurium provides limited prevention of muscular fibrillation due to succinylcholine, but the choice of dose often depends on user experience, and there have been no previous studies of age-related doses of cisatracurium for the prevention of muscular fibrillation caused by succinylcholine, and its half-effective amount (ED50) has not been established. In this study, patients treated with elective general anesthesia surgery were the subjects, and in the process of general anesthesia induction, cis-atracurium was pretreated to evaluate the degree of inhibition of muscular fibrillation caused by succinylcholine, and half of the effective dose of cis-atracurium inhibition of muscular fibrillation caused by succinylcholine was calculated by sequential method.

ELIGIBILITY:
Inclusion Criteria:

1. Ages ranged from 18 to 80.
2. ASA # or # level.

Exclusion Criteria:

* Allergy or contraindication to cisatracurium or succinylcholine;
* Associated with cardiovascular disease, diabetes, hyperkalemia, increased intraocular pressure, increased intracranial pressure, gastroesophageal reflux, difficult airway, malignant hyperthermia, neuromuscular disease Sick;
* Take drugs that may affect neuromuscular function before surgery
* Liver or kidney failure
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
The appearance of fasciculation Yes or No | an average of 2 minutes
  Yes or No
The levels of fasciculation | an average of 2 minutes
  Fasciculation after the administration of medications was examined and graded by an anesthesiologist using four-point Likert scale: Grade 0 = no fasciculation; Grade 1 = mild, fine fasciculations of the eyes, neck, face, or fingers, without limb movement; Grade 2 = moderate fasciculations occurring at more than two sites or obvious limb movement; and Grade 3 = vigorous or severe, sustained, and widespread fasciculations in the trunk and limbs.

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu, China